CLINICAL TRIAL: NCT01816087
Title: Study AGE - Part 2 (Active Geriatric Evaluation for General Practitioner), Performances of a Brief Assessment Tool for the Early Diagnosis of Geriatric Syndromes by Primary Care Physicians
Brief Title: Performances of a Brief Assessment Tool for the Early Diagnosis of Geriatric Syndromes by Primary Care Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Nicolas Senn, MD PhD, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 287/2012
Record Dates: First submitted 2013-02-20; First posted 2013-03-21 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Cognitive Impairment; Mood Disorders; Urinary Incontinence; Malnutrition; Osteoporosis; Hearing Impairment; Visual Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Mood Disorders; Urinary Incontinence; Malnutrition; Osteoporosis; Hearing Loss; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- brief assessment tool (BAT) (Experimental): all participants will have a brief assessment tool (BAT) for the identification of geriatric syndromes performed by their general practitioner. Afterwards, all participants will have a full geriatric assessment performed by geriatricians
  Interventions: Other: brief geriatric assessment

INTERVENTIONS:
Other: brief geriatric assessment — All participants will be screened for geriatric syndromes using the brief assessment tool. Mix a simple questions and simple tests

SUMMARY:
The AGE (Active Geriatric Evaluation) aims to develop a brief assessment tool adapted to the primary care setting.

DETAILED DESCRIPTION:
The AGE (Active Geriatric Evaluation) program is a collaborative project between a primary care institution and a specialised geriatric unit that aims to develop a brief assessment tool (BAT) adapted to the primary care setting. The objective of this study is to assess the performances of the BAT to identify major geriatric syndromes: cognitive impairment; mood disorder; functional impairment; urinary incontinence; malnutrition; gait and balance impairment; osteoporosis; hearing impairment; visual impairment.

In order to achieve our objective, we plan to recruit 155 patients > 70 years old in primary care settings for which primary care physicians will perform the BAT (composed of specific questions and clinical exams). At the end of the consultation, the primary care physician will fill a questionnaire where the absence/presence of syndromes will be recorded (according to the findings of the BAT). Each patient will be then seen a second time by expert geriatricians that will perform a full geriatric evaluation (90 minutes). This will allow to calculate the performances of the intervention (BAT) in terms of sensibility /specificity,...

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years
* follow-up by general practitioner
* good understanding of french or presence of a translater
* No previous or on-going geriatric consultation
* Patient able to provide consent or a relative is present that can provide a consent instead

Exclusion Criteria:

* Age < 70 years
* No follow-up by general practitioner
* Unable to understand French or absence of a translater
* On-going geriatric follow-up
* Patient unable to provide consent or a relative is absent

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sensibility and specificity | one year
  performances of the brief assessment tool (BAT) will be measured by calculating sensibility and specificity for each of the geriatric syndromes: cognitive impairment; mood disorder; functional impairment; urinary incontinence; malnutrition; gait and balance impairment; osteoporosis; hearing impairment; visual impairment

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Senn, MD PhD, Principal Investigator — Department of ambulatory care and community medicine, University of Lausanne, Switzerland
Locations (1):
- Departement of Ambulatory Care and Community Medicine, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Mueller YK, Monod S, Locatelli I, Bula C, Cornuz J, Senn N. Performance of a brief geriatric evaluation compared to a comprehensive geriatric assessment for detection of geriatric syndromes in family medicine: a prospective diagnostic study. BMC Geriatr. 2018 Mar 13;18(1):72. doi: 10.1186/s12877-018-0761-z. PMID 29534680